CLINICAL TRIAL: NCT00540098
Title: A Randomized, Controlled Trial on the Effects of Paroxetine Versus Placebo in Combination With Aerobic Exercise or Relaxation Training in the Treatment of Panic Disorder
Brief Title: Paroxetine vs Placebo Combined With Aerobic Exercise or Relaxation in Panic Disorder
Acronym: Exparox
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 290060/552
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Panic Disorder
Keywords: panic disorder; pharmacotherapy; non-pharmacological treatment; SSRI; paroxetine; exercise
MeSH Terms: conditions — Panic Disorder; Motor Activity | interventions — Paroxetine; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Paroxetine + aerobic exercise
  Interventions: Drug: paroxetine + aerobic exercise
- 2 (Active Comparator): Paroxetine + relaxation
  Interventions: Drug: Paroxetine + relaxation
- 3 (Active Comparator): Placebo + aerobic exercise
  Interventions: Drug: Placebo + aerobic exercise
- 4 (Placebo Comparator): Placebo + relaxation
  Interventions: Drug: Placebo + relaxation

INTERVENTIONS:
Drug: paroxetine + aerobic exercise — paroxetine, 40 mg once daily + regular aerobic exercise
  Arms: 1
Drug: Paroxetine + relaxation — paroxetine, 40 mg once daily + regular relaxation training
  Arms: 2
Drug: Placebo + aerobic exercise — placebo pill once daily + regular aerobic exercise
  Arms: 3
Drug: Placebo + relaxation — placebo pill once daily + regular relaxation training
  Arms: 4

SUMMARY:
Efficacy and safety of a 10-weeks treatment protocol of paroxetine vs. placebo in combination with regular aerobic exercise (running) or regular relaxation training in the treatment of panic disorder.

DETAILED DESCRIPTION:
In continuation of prior work from our group (Broocks A, Bandelow B, Pekrun G, et al. Comparison of aerobic exercise, clomipramine, and placebo in the treatment of panic disorder. Am J Psychiatry 1998; 155(5):603-9.) it is the purpose of this trial to test the assumed superiority of a combined therapy of paroxetine and aerobic exercise compared to placebo or unspecific relaxation training in panic disorder. Participants were randomized to a 10 week treatment protocol of paroxetine 40 mg daily or placebo in combination with regular exercise or regular relaxation after having given informed consent and screening of in- and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Panic disorder with or without agoraphobia due to DSM-IV
* Written informed consent
* Score of 17 or more on the P&A scale
* Score on the CGI of 4 or more (markedly ill)

Exclusion Criteria:

* Pregnancy, lactating or insufficient contraception (pearl index >1)
* Other psychiatric disorders such as psychoses, addictive disorders, dementia, etc.
* Clinically relevant abnormalities in physical examination or laboratory results
* Prior major depression or bipolar disorder
* Suicidality
* psychotropic medication other than promethazine
* current psychological treatment
* unable to perform regular aerobic exercise

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2001-09; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Severity of Panic disorder due to Scores on the Panic and Agoraphobia Scale (P&A) | Baseline to endpoint (10 weeks)
Severity of panic disorder due to scores on the Clinical Global Impression scale (CGI) | Baseline to endpoint (10 weeks)

SECONDARY OUTCOMES:
Symptom severity due to Hamilton Anxiety Scale (HAMA) | Baseline to endpoint (10 weeks)
Symptom severity due to the Montgomery and Asberg depression rating scale (MADRS) | Baseline to endpoint (10 weeks)
Response and remission analysis between groups | LOCF-analysis

CONTACTS AND LOCATIONS:
Overall Officials: Borwin Bandelow, Prof, MD, Principal Investigator — University of Göttingen
Locations (1):
- University of Göttingen, Dept of Psychiatry and Psychotherapy, Göttingen, Germany

REFERENCES:
- [Background] Broocks A, Bandelow B, Pekrun G, George A, Meyer T, Bartmann U, Hillmer-Vogel U, Ruther E. Comparison of aerobic exercise, clomipramine, and placebo in the treatment of panic disorder. Am J Psychiatry. 1998 May;155(5):603-9. doi: 10.1176/ajp.155.5.603. PMID 9585709